CLINICAL TRIAL: NCT01745042
Title: Impact of Fat Distribution on Metabolic, Cardiovascular and Symptomatic Aspects in Postmenopausal Women
Brief Title: Anthropometric, Metabolic, Cardiovascular and Symptomatic Profile in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Fernanda Rossi Paolillo, Federal University of São Carlos, University of Sao Paulo
Other Study IDs: 150949/2011-1
Record Dates: First submitted 2012-12-03; First posted 2012-12-07 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Postmenopausal Disorder
Keywords: Postmenopausal Women; Body Composition; Metabolic Syndrome; Menopause Symptoms
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- android postmenopausal women: Clinical exams
  Interventions: Other: Clinical exams
- gynoid postmenopausal women: Clinical exams
  Interventions: Other: Clinical exams

INTERVENTIONS:
Other: Clinical exams — Physiological and biochemical tests; quality of life questionnaire; body composition measurement

SUMMARY:
The purpose of this study is to investigate anthropometric, metabolic, cardiovascular and symptomatic profiles in postmenopausal women.

DETAILED DESCRIPTION:
When aging, the body composition changes, leading to a reduction of muscle mass and strength, and to an increase in total body fat. These body composition changes have especially been observed in postmenopausal women, due to the hormonal changes taking place. After the menopause, the gynoid fat distribution with fat deposits in the gluteo-femoral region changes to an android fat distribution with an increased upper body fat, especially in the abdominal region. These consequences of the menopause associated with a decrease in aerobic capacity and reduced total energy expenditure may lead to the metabolic syndrome (MetS). The aim of this study was to investigate the anthropometric, metabolic, cardiovascular and symptomatic profile in gynoid and android postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Caucasian
* 50-60 years of age

Exclusion Criteria:

* Neurological disease
* Pulmonary disease
* Cardiac disease
* Oncological disease
* Musculotendinous or articular injuries
* Hormone replacement therapy
* Cigarette smoking

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Postmenopausal women from a community sample of São Carlos city - São Paulo State - Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Relationships between postmenopause and fat distribution | Baseline
  Anthropometric measurements: waist-to-hip ratio and body mass index

SECONDARY OUTCOMES:
Comparison of aerobic capacity between android and gynoid postmenopausal women | Baseline
  Progressive aerobic testing on treadmill (Modified Bruce Protocol): estimated maximum oxygen consumption; metabolic equivalents; blood pressure; heart rate
Comparison of metabolic parameters between android and gynoid postmenopausal women | Baseline
  Biochemical tests: the serum level of estradiol, urea, creatinine, triglycerides, total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, very low-density lipoprotein (VLDL) cholesterol, insulin and glucose
Comparison of quality of life between android and gynoid postmenopausal women | Baseline
  Menopause Rating Scale (MRS): somatic symptoms; psychological symptoms; urogenital-sexual problems
Comparison of the body composition between android and gynoid postmenopausal women | Baseline
  Body composition: bipolar electrical bioimpedance (body fat and lean mass) and skinfolds (triceps, subscapular, suprailiac, abdominal, anterior thigh, medial calf)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Borghi-Silva, Ph.D, Study Director — Department of Physical Therapy, Federal University of São Carlos (UFSCar); Cristina Kurachi, Ph.D, Study Director — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Vanderlei S Bagnato, Ph.D, Study Director — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Fernanda R. Paolillo, Ph.D, Principal Investigator — Physics Institute of São Carlos (IFSC), University of São Paulo (USP)
Locations (1):
- Optics Group from Physics Institute of São Carlos (IFSC), University of São Paulo (USP), São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Paolillo FR, Milan JC, Bueno Pde G, Paolillo AR, Borghi-Silva A, Parizotto NA, Arena R, Kurachi C, Bagnato VS. Effects of excess body mass on strength and fatigability of quadriceps in postmenopausal women. Menopause. 2012 May;19(5):556-61. doi: 10.1097/gme.0b013e3182364e80. PMID 22089183
- [Background] Paolillo FR, Milan JC, Aniceto IV, Barreto SG, Rebelatto JR, Borghi-Silva A, Parizotto NA, Kurachi C, Bagnato VS. Effects of infrared-LED illumination applied during high-intensity treadmill training in postmenopausal women. Photomed Laser Surg. 2011 Sep;29(9):639-45. doi: 10.1089/pho.2010.2961. Epub 2011 Jul 12. PMID 21749263
- [Background] Paolillo FR, Corazza AV, Borghi-Silva A, Parizotto NA, Kurachi C, Bagnato VS. Infrared LED irradiation applied during high-intensity treadmill training improves maximal exercise tolerance in postmenopausal women: a 6-month longitudinal study. Lasers Med Sci. 2013 Feb;28(2):415-22. doi: 10.1007/s10103-012-1062-y. Epub 2012 Mar 2. PMID 22382875
- [Background] Blumel JE, Legorreta D, Chedraui P, Ayala F, Bencosme A, Danckers L, Lange D, Espinoza MT, Gomez G, Grandia E, Izaguirre H, Manriquez V, Martino M, Navarro D, Ojeda E, Onatra W, Pozzo E, Prada M, Royer M, Saavedra JM, Sayegh F, Tserotas K, Vallejo MS, Zuniga C; Collaborative Group for Research of the Climacteric in Latin America (REDLINC). Optimal waist circumference cutoff value for defining the metabolic syndrome in postmenopausal Latin American women. Menopause. 2012 Apr;19(4):433-7. doi: 10.1097/gme.0b013e318231fc79. PMID 22067278
- [Background] Despres JP, Lemieux I. Abdominal obesity and metabolic syndrome. Nature. 2006 Dec 14;444(7121):881-7. doi: 10.1038/nature05488. PMID 17167477